CLINICAL TRIAL: NCT04867824
Title: Comparison of Lavender vs Vanilla Essential Oil as Complementary Analgesia for Frenotomy in Healthy Newborns: a Randomized Clinical Trial.
Brief Title: The Use of Lavender vs Vanilla Essential Oil as Complementary Analgesia for Frenotomy in Healthy Newborns
Acronym: LVEO-SME1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021/9731/I
Record Dates: First submitted 2021-04-27; First posted 2021-04-30 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Ankyloglossia
Keywords: ankyloglossia; tongue-tie; aromatherapy; lavender; vanilla; pain; neonate; frenotomy
MeSH Terms: conditions — Ankyloglossia; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): The neonate will be taken to the neonatal unit and monitored with a pulse-oximeter before, during and after the procedure. We will swaddle it, will administer 1 mL of oral sucrose, let the newborn suck for 2 minutes prior to the procedure, and will have a 7 x 7 cm gauze pad with 1 drop of 100% pure LEO (Pranarôm España S.L.) placed 2 cm under the nose for 2 minutes prior to starting the frenotomy and during the procedure.
  Interventions: Dietary Supplement: Control (use of inhaled lavender essential oil)
- Case (Experimental): The neonate will be taken to the neonatal unit and monitored with a pulse-oximeter before, during and after the procedure. We will swaddle it, will administer 1 mL of oral sucrose, let the newborn suck for 2 minutes prior to the procedure, and will have a 7 x 7 cm gauze pad with 1 drop of 100% pure vanilla essential oil (Pranarôm España S.L.) placed 2 cm under the nose for 2 minutes prior to starting the frenotomy and during the procedure.
  Interventions: Dietary Supplement: Case (use of inhaled vanilla essential oil)

INTERVENTIONS:
Dietary Supplement: Case (use of inhaled vanilla essential oil) — Use of inhaled vanilla essential oil during frenotomy for a tongue-tie
  Arms: Case
Dietary Supplement: Control (use of inhaled lavender essential oil) — Use of inhaled lavender essential oil during frenotomy for a tongue-tie
  Arms: Control

SUMMARY:
Clipping of the tongue-tie is a common procedure that physicians perform in our neonatal unit to help establish breastfeeding. It is a painful technique where the measures usually performed to control pain (such as sucking) cannot be done at the time of the clipping because the technique is performed on the tongue. A previous study conducted at our center proved the benefits of inhaled lavender essential oil to control pain during frenotomy, for which inhaled essential oil is now routinely used when clipping a tongue-tie. The aim of this study was to compare the analgesic/soothing effect of inhaled lavender essential oil vs inhaled vanilla essential oil during the clipping of the tongue-tie. Participants will be newborns born at our hospital during the study period (expected to be May to December 2021). Patients will be offered to participate and will be enrolled in the study if their parents agree to and sign an informed consent. The use of inhaled lavender and vanilla essential oils is safe. No side effects have been found with their use. The procedure of the frenotomy will not change for patients who are enrolled in the study. At the moment, inhaled lavender essential oil is used as complementary analgesia for the clipping of tongue-ties in our neonatal unit. By demonstrating which of the two oils has better results, the investigators aim to improve pain management of the patients who undergo a frenotomy. This study will take place at the neonatal unit of Hospital del Mar, Barcelona, Spain.

DETAILED DESCRIPTION:
A randomized clinical trial will be conducted with the neonates born at our hospital or less than 15 days old who undergo a frenotomy for type 3 tongue-ties according to Coryllos classification and the Hazelbaker tool during the study period (expected to take place from May to December 2021). Pain will be assessed by means of crying time, the highest Neonatal Infant Pain Scale (NIPS) score in the five minutes post procedure, increase in heart rate (HR) and decrease in oxygen saturation (satO2) pre/post-procedure. NIPS evaluates facial expression, crying, breathing pattern, arm and leg position, and state of arousal on a scale from 0 to 7, where 0-2 means no pain to mild pain, 3-4 mild to moderate pain, and >4 severe pain. In an exploratory preliminary study prior to the intervention, a mean (SD) crying time of 19.80 (21.14) seconds was observed. In order to detect a difference of 10 seconds in crying time, the investigators calculated that a sample size of 71 patients per group would be required in order to draw conclusions with a CI 95% and a power of 80%. Patients will be enrolled if their parents agree to and sign a written informed consent. Demographic (sex, gestational age, birth weight, age in hours at the time of frenotomy) and clinical variables (HR and satO2 before, during, and after the procedure, whether there is crying or not during the procedure, length of crying time in seconds, presence of side effects during the procedure (apnea, desaturation, others) and highest NIPS score within the first 5 minutes after the procedure) will be recorded. The independent variable will be the use of inhaled lavender essential oil (LEO) or the use of inhaled vanilla essential oil during frenotomy. The dependent variables will be: HR and satO2 pre and post procedure, presence of crying and duration, hours of life at the time of the frenotomy, and the NIPS score. The controlled variables will be: gestational age, sex, and birth weight.

Healthcare providers assess for the presence of ankyloglossia as part of the routine neonatal evaluation and offer a frenotomy to all tongue-tied patients. The examiner grades the ankyloglossia based on Coryllos's criteria and the Hazelbaker tool to assess its impact on tongue movement and on breastfeeding. A lingual frenulum is symptomatic if it scores 8 points or less in appearance and/or 11 points or less in function according to Hazelbaker. Advice and help with positioning and attachment for breastfeeding is provided to all the mothers by IBCLC (International Board Certified Lactation Consultant) nurses. During the study period, if a patient with a type 3 tongue-tie is identified, the patient's parents will be offered to participate in this study. Accepted patients will be allocated into case (vanilla essential oil) or control (LEO) group by simple random sampling using the program OxMAR (Online Minimization and Randomization for Clinical Trials).

During the frenotomy the neonate will be taken to the neonatal unit and monitored with a pulse-oximeter (COVIDIEN Nellcor Portable SpO2 Patient Monitoring System PM10N, Covidien Ireland Limited, IDA Business & Technology Park, Tullamore, Ireland) before, during and after the procedure. For both groups the neonates will de swaddled, administered 1 mL of oral sucrose, and allowed to suck for 2 minutes prior to the procedure. The control group will have a 7 x 7 cm gauze pad with 1 drop of 100% pure LEO (Pranarôm España S.L.) placed 2 cm under their nose for 2 minutes prior to starting the frenotomy and during the procedure. The case group will have a 7 x 7 cm gauze pad with 1 drop of 100% pure vanilla essential oil (Pranarôm España S.L.) placed 2 cm under their nose for 2 minutes prior to starting the frenotomy and during the procedure. The bottle of both essential oils has a dropper that always dispenses the same amount of oil per drop. The procedure will not start until the patient is calm and has a NIPS score of 0. Frenotomy will be performed by one of the three staff neonatologists using Coryllos' technique: placing a sterile groove director under the tongue straddling the frenulum, holding the frenulum in place with visualization of tongue base and frenulum, and snipping the frenulum with a scissor along the underside of the tongue to its base just proximal to the genioglossus muscle, until a full release is achieved. Once the procedure is completed, the gauze pad will be removed and vital signs recorded, as well as whether the baby cried or not, the seconds crying lasted, and the post procedure NIPS score on a data collection sheet. If a neonate cries, calming techniques such as holding, swaddling, and sucking will be employed. Following the frenotomy, the neonate will be returned to the mother for breastfeeding.

Statistical analysis: Quantitative variables (gestational age, birth weight, age at frenotomy, heart rate pre and post-procedure, increase in heart rate postprocedure, oxygen saturation pre and post-procedure, decrease in oxygen saturation post-procedure, and duration of crying) will be described using the mean, standard deviation, and 95% confidence interval (CI); case vs control groups will be compared with a Student's t test. Sex, the presence of crying, and adverse effects between the two groups will be presented in percentages and will be compared using Fisher's exact test. NIPS scores between cases and controls will be compared with the Wilcoxon rank-sum (Mann-Whitney) test. Statistical significance will be set for a p <0.05. To perform statistical analyses, the investigators will use STATA version 15.1 (StataCorp, College Station, TX, USA).

Our hospital Ethics Committee (CEIm-PSMAR) will approve this study (reference code: 2021/9731/I). Prior to patient enrollment, the investigators will obtain a signed informed consent from the neonate's parents. This study will be conducted according to the ethics code of the Barcelona Medical Association and the principles of the Helsinki-Fortaleza Declaration 2013.

ELIGIBILITY:
Inclusion Criteria:

* Healthy full-term neonates born at Hospital del Mar (Barcelona, Spain), or less than 15 days old who had been discharged and returned for the frenotomy, who underwent a frenotomy for type 3 tongue-ties according to Coryllos classification and the Hazelbaker tool during the study period

Exclusion Criteria:

* Refusal of the patient's parents to participate

Ages: 0 Days to 15 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 142 (Estimated)
Dates: Start 2021-05-10 (Estimated); Primary Completion 2021-12-09 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Crying length | Up to 5 minutes post-procedure
  Crying length after the frenotomy in seconds
NIPS score | Up to 5 minutes post-procedure
  Neonatal Infant Pain Score value (0-7). NIPS evaluates facial expression, crying, breathing pattern, arm and leg position, and state of arousal on a scale from 0 to 7, where 0-2 means no pain to mild pain, 3-4 mild to moderate pain, and >4 severe pain.
Increase in heart rate | Up to 5 minutes post-procedure
  Increase in heart rate pre/post-procedure (beats per minute)
Decrease in oxygen saturation | Up to 5 minutes post-procedure
  Decrease in oxygen saturation (%)

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Maya-Enero, Ph.D., M.D., Principal Investigator — Hospital del Mar

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goubet N, Strasbaugh K, Chesney J. Familiarity breeds content? Soothing effect of a familiar odor on full-term newborns. J Dev Behav Pediatr. 2007 Jun;28(3):189-94. doi: 10.1097/dbp.0b013e31802d0b8d. PMID 17565285
- [Background] Johnston CC, Fernandes AM, Campbell-Yeo M. Pain in neonates is different. Pain. 2011 Mar;152(3 Suppl):S65-S73. doi: 10.1016/j.pain.2010.10.008. Epub 2010 Oct 23. PMID 20971562
- [Background] Fitri SYR, Wardhani V, Rakhmawati W, Pahria T, Hendrawati S. Culturally Based Practice in Neonatal Procedural Pain Management: A Mini Review. Front Pediatr. 2020 Sep 3;8:540. doi: 10.3389/fped.2020.00540. eCollection 2020. PMID 33014934
- [Background] Razaghi N, Aemmi SZ, Sadat Hoseini AS, Boskabadi H, Mohebbi T, Ramezani M. The effectiveness of familiar olfactory stimulation with lavender scent and glucose on the pain of blood sampling in term neonates: A randomized controlled clinical trial. Complement Ther Med. 2020 Mar;49:102289. doi: 10.1016/j.ctim.2019.102289. Epub 2019 Dec 26. PMID 32147068
- [Background] Mitchell A, Boss BJ. Adverse effects of pain on the nervous systems of newborns and young children: a review of the literature. J Neurosci Nurs. 2002 Oct;34(5):228-36. doi: 10.1097/01376517-200210000-00002. PMID 12391738
- [Background] Stevens B, Yamada J, Ohlsson A, Haliburton S, Shorkey A. Sucrose for analgesia in newborn infants undergoing painful procedures. Cochrane Database Syst Rev. 2016 Jul 16;7(7):CD001069. doi: 10.1002/14651858.CD001069.pub5. PMID 27420164
- [Background] Harrison D, Larocque C, Bueno M, Stokes Y, Turner L, Hutton B, Stevens B. Sweet Solutions to Reduce Procedural Pain in Neonates: A Meta-analysis. Pediatrics. 2017 Jan;139(1):e20160955. doi: 10.1542/peds.2016-0955. Epub 2016 Dec 16. PMID 27986905
- [Background] Leng HY, Zheng XL, Yan L, Zhang XH, He HY, Xiang M. [Effects of different types and concentration of oral sweet solution on reducing neonatal pain during heel lance procedures]. Zhonghua Er Ke Za Zhi. 2013 Sep;51(9):654-8. Chinese. PMID 24330983
- [Background] Jones JE, Kassity N. Varieties of alternative experience: complementary care in the neonatal intensive care unit. Clin Obstet Gynecol. 2001 Dec;44(4):750-68. doi: 10.1097/00003081-200112000-00012. No abstract available. PMID 11600855
- [Background] Akcan E, Polat S. Comparative Effect of the Smells of Amniotic Fluid, Breast Milk, and Lavender on Newborns' Pain During Heel Lance. Breastfeed Med. 2016 Aug;11(6):309-314. doi: 10.1089/bfm.2015.0174. Epub 2016 Jun 17. PMID 27315487
- [Background] Vaziri F, Khosropoor M, Hidari M, Pourahmad S, Morshed Behbahani B, Saki F. The Effect of Aromatherapy by Lavender Oil on Infant Vaccination Pain: a Double Blind Randomized Controlled Trial. J Caring Sci. 2019 Mar 1;8(1):17-21. doi: 10.15171/jcs.2019.003. eCollection 2019 Mar. PMID 30915309
- [Background] Maya-Enero S, Perez-Perez M, Ruiz-Guzman L, Duran-Jorda X, Lopez-Vilchez MA. Prevalence of neonatal ankyloglossia in a tertiary care hospital in Spain: a transversal cross-sectional study. Eur J Pediatr. 2021 Mar;180(3):751-757. doi: 10.1007/s00431-020-03781-7. Epub 2020 Aug 15. PMID 32803423
- [Background] Cetinkaya B, Basbakkal Z. The effectiveness of aromatherapy massage using lavender oil as a treatment for infantile colic. Int J Nurs Pract. 2012 Apr;18(2):164-9. doi: 10.1111/j.1440-172X.2012.02015.x. PMID 22435980
- [Background] Field T, Field T, Cullen C, Largie S, Diego M, Schanberg S, Kuhn C. Lavender bath oil reduces stress and crying and enhances sleep in very young infants. Early Hum Dev. 2008 Jun;84(6):399-401. doi: 10.1016/j.earlhumdev.2007.10.008. Epub 2007 Nov 28. PMID 18053656
- [Background] Lawrence J, Alcock D, McGrath P, Kay J, MacMurray SB, Dulberg C. The development of a tool to assess neonatal pain. Neonatal Netw. 1993 Sep;12(6):59-66. PMID 8413140
- [Background] Lopez V, Nielsen B, Solas M, Ramirez MJ, Jager AK. Exploring Pharmacological Mechanisms of Lavender (Lavandula angustifolia) Essential Oil on Central Nervous System Targets. Front Pharmacol. 2017 May 19;8:280. doi: 10.3389/fphar.2017.00280. eCollection 2017. PMID 28579958
- [Background] Habanananda T. Non-pharmacological pain relief in labour. J Med Assoc Thai. 2004 Oct;87 Suppl 3:S194-202. PMID 21213523
- [Background] Goubet N, Rattaz C, Pierrat V, Bullinger A, Lequien P. Olfactory experience mediates response to pain in preterm newborns. Dev Psychobiol. 2003 Mar;42(2):171-80. doi: 10.1002/dev.10085. PMID 12555281
- [Background] Sadathosseini AS, Negarandeh R, Movahedi Z. The effect of a familiar scent on the behavioral and physiological pain responses in neonates. Pain Manag Nurs. 2013 Dec;14(4):e196-e203. doi: 10.1016/j.pmn.2011.10.003. Epub 2012 Feb 28. PMID 24315273
- [Background] Mikami-Saito Y, Maekawa M, Wada Y, Kanno T, Kurihara A, Sato Y, Yamamoto T, Arai-Ichinoi N, Kure S. Essential oils can cause false-positive results of medium-chain acyl-CoA dehydrogenase deficiency. Mol Genet Metab Rep. 2020 Nov 5;25:100674. doi: 10.1016/j.ymgmr.2020.100674. eCollection 2020 Dec. PMID 33204637
- [Derived] Maya-Enero S, Fabregas-Mitjans M, Llufriu-Marques RM, Candel-Pau J, Garcia-Garcia J, Lopez-Vilchez MA. Comparison of the analgesic effect of inhaled lavender vs vanilla essential oil for neonatal frenotomy: a randomized clinical trial (NCT04867824). Eur J Pediatr. 2022 Nov;181(11):3923-3929. doi: 10.1007/s00431-022-04608-3. Epub 2022 Sep 8. PMID 36076107